CLINICAL TRIAL: NCT05086952
Title: Pivotal Relative Bioavailability Study to Investigate the Pharmacokinetics and Food Effect of Single Oral Doses of Vericiguat Given as Pediatric Oral Suspension Formulations in Comparison to the 10 mg IR Tablet in Healthy Male Participants in a Randomized, Open-label, 4-fold Crossover Design
Brief Title: A Study in Healthy Adult Male Participants to Learn the Way Vericiguat is Absorbed With and Without Food When Taken as a Single Dose in Liquid Form Suitable for Children Compared to a 10 Milligram (mg) Tablet That Releases the Active Substance Immediately
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 21150; 2021-001199-40 (EudraCT Number)
Record Dates: First submitted 2021-10-01; First posted 2021-10-21 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure; Children
MeSH Terms: conditions — Heart Failure | interventions — vericiguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- B-A-D-C (Experimental): 4-fold crossover design with 4 interventions, 4 intervention periods, and 4 intervention sequences. (according to Williams design [balanced for 1-period-carry-over]).
  Interventions: Drug: Vericiguat (BAY1021189) - Intervention A; Drug: Vericiguat (BAY1021189) - Intervention B; Drug: Vericiguat (BAY1021189) - Intervention C; Drug: Vericiguat (Verquvo, BAY1021189) - Intervention D
- C-D-A-B (Experimental): 4-fold crossover design with 4 interventions, 4 intervention periods, and 4 intervention sequences. (according to Williams design [balanced for 1-period-carry-over]).
  Interventions: Drug: Vericiguat (BAY1021189) - Intervention A; Drug: Vericiguat (BAY1021189) - Intervention B; Drug: Vericiguat (BAY1021189) - Intervention C; Drug: Vericiguat (Verquvo, BAY1021189) - Intervention D
- D-B-C-A (Experimental): 4-fold crossover design with 4 interventions, 4 intervention periods, and 4 intervention sequences. (according to Williams design [balanced for 1-period-carry-over]).
  Interventions: Drug: Vericiguat (BAY1021189) - Intervention A; Drug: Vericiguat (BAY1021189) - Intervention B; Drug: Vericiguat (BAY1021189) - Intervention C; Drug: Vericiguat (Verquvo, BAY1021189) - Intervention D
- A-C-B-D (Experimental): 4-fold crossover design with 4 interventions, 4 intervention periods, and 4 intervention sequences. (according to Williams design [balanced for 1-period-carry-over]).
  Interventions: Drug: Vericiguat (BAY1021189) - Intervention A; Drug: Vericiguat (BAY1021189) - Intervention B; Drug: Vericiguat (BAY1021189) - Intervention C; Drug: Vericiguat (Verquvo, BAY1021189) - Intervention D

INTERVENTIONS:
Drug: Vericiguat (BAY1021189) - Intervention A — Single dose of 10 mg vericiguat high-concentration pediatric formulation (oral liquid formulation) in fed state.
Drug: Vericiguat (BAY1021189) - Intervention B — Single dose of 10 mg vericiguat high-concentration pediatric formulation (oral liquid formulation) in fasted state.
Drug: Vericiguat (BAY1021189) - Intervention C — Single dose of 2.5 mg vericiguat low-concentration pediatric formulation (oral liquid formulation) in fed state.
Drug: Vericiguat (Verquvo, BAY1021189) - Intervention D — Single dose of 10 mg vericiguat immediate release (IR) intact tablet in fed state.

SUMMARY:
Researchers are looking for a better way to treat heart failure, a condition in which the heart does not pump blood as well as it should. Heart failure can happen in both adults and children.

The study treatment, vericiguat, is already available for doctors to give to adults who have heart failure. It works by increasing the activity of an enzyme called soluble guanylate cyclase (sGC). The sGC enzyme helps regulate the heart and blood circulation.

The current form of vericiguat is a tablet that releases the "active substance" immediately. The "active substance" is the part of the drug that works in the body to treat the condition. Vericiguat is currently only available as a treatment for adults. Researchers think vericiguat could help treat children with heart failure, but think it will be easiest for them to take a liquid treatment.

Another study is planned to find out how well vericiguat works in children who have a specific type of heart failure. Before researchers can give vericiguat to children, they must first study different doses and ways of taking vericiguat in adults. In this study, the researchers will study a new liquid form of vericiguat in adults. This form is also known as the "pediatric formulation".

In this study, the researchers want to find out how the new pediatric formulation of vericiguat moves into, through, and out of the body compared to the currently approved tablet form for adults. The researchers also want to find out if eating food affects the new pediatric formulation differently than the current tablet form of vericiguat.

The study will include about 36 healthy white male participants aged between 18 and 45 years old.

During this study, the participants will all take 4 different treatments in different orders. They will take:

* a high dose of vericiguat in the new pediatric formulation, with food
* a high dose of vericiguat in the new pediatric formulation, without food
* a low dose of vericiguat in the new pediatric formulation, with food
* a dose of the currently available tablet form, with food While taking each study treatment, the participants will stay at the study site for 4 days. There will be a break of at least 10 days between each treatment. Overall, the participants will be in this study for about 11 weeks.

During the study, the participants will:

* have blood and urine samples taken
* have their overall health and heart health checked
* answer questions about how the new pediatric formulation tastes
* answer questions about any adverse events they are having An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if they do not think the adverse events might be related to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* Age 18 -45 years
* Body Mass Index (BMI): above or equal 18.5 and below or equal 29.9 kg / m²

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Febrile illness (temperature ≥38.0 oC) within 4 weeks prior to admission to the ward
* A history of relevant diseases of vital organs, of the central nervous system or other organs
* A history of relevant smell and / or taste disorders
* Relevant diseases within the last 4 weeks prior to the first study intervention administration
* Known gastro-intestinal disorders (e.g. stomach ulcers, duodenal ulcers, gastro-intestinal bleeding) or inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis)
* Regular use of medicines in the 4 weeks prior to first dosing
* Regular use of therapeutic or recreational drugs (e.g. carnitine products, anabolics, high-dose vitamins)
* Use of medication (prescription or over the counter) or herbal products within 2 weeks before first study intervention administration which could oppose the study objectives or which might influence them
* Criteria which in the opinion of the investigator preclude participation for scientific reasons, for reasons of compliance, or for reasons of the participant's safety

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
AUC of vericiguat (a single oral dose of the pediatric high concentration formulation in comparison to vericiguat intact tablet in fed condition) | From pre-dose until 72 hours after dosing in each intervention period
  AUC: area under the concentration vs. time curve from zero to infinity after single (first) dose, calculated up by linear trapezoidal rule, down by logarithmic trapezoidal rule
AUC(0-tlast) of vericiguat (a single oral dose of the pediatric high concentration formulation in comparison to vericiguat intact tablet in fed condition) | From pre-dose until 72 hours after dosing in each intervention period
  AUC(0-tlast): AUC from time 0 to the last data point > lower limit of quantitation (LLOQ)
Cmax of vericiguat (a single oral dose of the pediatric high concentration formulation in comparison to vericiguat intact tablet in fed condition) | From pre-dose until 72 hours after dosing in each intervention period
  Cmax: maximum observed drug concentration in measured matrix after single dose administration

SECONDARY OUTCOMES:
AUC/D of vericiguat ( a single oral dose of 2.5 mg of the pediatric low-concentration formulation in comparison to 10 mg vericiguat intact tablet in fed condition) | From pre-dose until 72 hours after dosing in each intervention period
  AUC/D: AUC divided by dose
AUC(0-tlast)/D of vericiguat ( a single oral dose of 2.5 mg of the pediatric low-concentration formulation in comparison to 10 mg vericiguat intact tablet in fed condition) | From pre-dose until 72 hours after dosing in each intervention period
  AUC(0-tlast)/D: AUC from time 0 to the last data point divided by dose
Cmax/D of vericiguat ( a single oral dose of 2.5 mg of the pediatric low-concentration formulation in comparison to 10 mg vericiguat intact tablet in fed condition) | From pre-dose until 72 hours after dosing in each intervention period
  Cmax/D: Cmax divided by dose
AUC/D of vericiguat (a single oral dose of 10 mg of the pediatric high-concentration formulation in comparison to a single oral dose of 2.5 mg of the pediatric low-concentration formulation in fed condition) | From pre-dose until 72 hours after dosing in each intervention period
AUC(0-tlast)/D of vericiguat (a single oral dose of 10 mg of the pediatric high-concentration formulation in comparison to a single oral dose of 2.5 mg of the pediatric low-concentration formulation in fed condition) | From pre-dose until 72 hours after dosing in each intervention period
Cmax/D of vericiguat (a single oral dose of 10 mg of the pediatric high-concentration formulation in comparison to a single oral dose of 2.5 mg of the pediatric low-concentration formulation in fed condition) | From pre-dose until 72 hours after dosing in each intervention period
Number of participants with treatment emergent adverse events (TEAEs) | From dosing to 5 days after each dose per period (estimate duration is 20 days)
Questionnaire by means of descriptive statistics | 0 - 30 minutes
  Questionnaire to assess the taste, smell, and appearance of the newly developed pediatric formulation of vericiguat.
AUC of vericiguat (a high fat, high calorie meal on the PK of vericiguat after a single oral dose of high-concentration pediatric formulation in comparison to the fasted state) | From pre-dose until 72 hours after dosing in each intervention period
AUC(0-tlast) of vericiguat (a high fat, high calorie meal on the PK of vericiguat after a single oral dose of high-concentration pediatric formulation in comparison to the fasted state) | From pre-dose until 72 hours after dosing in each intervention period
Cmax of vericiguat (a high fat, high calorie meal on the PK of vericiguat after a single oral dose of high-concentration pediatric formulation in comparison to the fasted state) | From pre-dose until 72 hours after dosing in each intervention period

CONTACTS AND LOCATIONS:
Locations (1):
- SocraTec R&D GmbH, Erfurt, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com